CLINICAL TRIAL: NCT00883077
Title: Combined Assessment of Colonic Permeability by Real Time Confocal Laser Endomicroscopy and Sucralose Absorption Test
Brief Title: Assessment of Colonic Permeability by Confocal Laser Endomicroscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Yan-Qing Li, Department of Gastroenterology, Qilu Hospital, Shandong University
Other Study IDs: 2009SDU-QILU-G01
Record Dates: First submitted 2009-04-15; First posted 2009-04-17 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Inflammatory Bowel Disease; Ulcerative Colitis; Irritable Bowel Syndrome
Keywords: permeability; inflammatory bowel disease; confocal laser endomicroscopy; irritable bowel syndrome
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsies during colonoscopy.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Inflammation: Patients with long standing history or short onset of ulcerative colitis.
- Healthy controls: Asymptomatic individuals admitted for health surveillance or patients for follow up after polypectomy.
- Irritable bowel syndrome: Patients admitted to outpatient department with symptoms meeting ROME III criteria of irritable bowel syndrome.

SUMMARY:
The purpose of this study is to evaluate the efficacy of confocal laser endomicroscopy in assessment of colonic permeability against conventional sugar absorption test.

DETAILED DESCRIPTION:
Increased intestinal permeability has been shown significant in many gastrointestinal diseases, including inflammatory bowel disease and recently irritable bowel syndrome. The conventional test methods of permeability is sugar absorption test which is neither reliable and practical. Confocal laser endomicrosopy is a newly developed device which allows in vivo and real time observation of gastrointestinal mucosa. In our preliminary study we found that the commonly used contrast agent, fluorescein sodium shew differences of leakage into colonic crypt lumen among different patients. The fluorescein leakage might be due to abnormal colonic permeability, so we planed to compare the fluorescein leakage under confocal laser endomicroscopy with conventional sucralose absorption test.

ELIGIBILITY:
Inclusion Criteria:

* Patients with history of ulcerative colitis
* Bowel habits alterations meeting IBS diagnosis criteria and indications for colonoscopy investigation
* Asymptomatic individuals for health surveillance or patients for follow up after polypectomy
* Patients complained of hemafecia but colonoscopy revealed only haemorrhoid

Exclusion Criteria:

* Known cancers or abdominal surgery
* Scheduled for endoscopic treatment
* Alarm symptoms such as anaemia, gastrointestinal bleeding or obstruction, marked weight loss, abdominal mass
* Under conditions such as:

  * ascites
  * jaundice
  * liver cirrhosis
  * impaired renal function
  * coagulopathy
  * fever
  * pregnancy
  * breastfeeding
* Inability to provide informed consent
* Known allergy to fluorescein sodium

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with indications for colonoscopy in Qilu Hospital outpatient and inpatient department are the study population of this study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-11 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Fluorescein leakage under confocal laser endomicroscopy observation of colonic mucosa. | Within the 30 minutes after injection of fluorescein

SECONDARY OUTCOMES:
Total sucralose excretion. | Within the 24 hours after drinking of sucralose

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PhD. MD., Study Director — Department of Gastroenterology, Qilu Hospital, Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China